CLINICAL TRIAL: NCT02000713
Title: Cervical Spinal Cord Metabolism and Microstructure in Amyotrophic Lateral Sclerosis(ALS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle Investigator was unable to fulfill responsibilities.
Sponsor: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00069508
Record Dates: First submitted 2013-11-08; First posted 2013-12-04 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Amyotrophic Lateral Sclerosis (Experimental): All subjects will be interviewed and administered a brief questionnaire to determine current disease severity. A brief neurological examination will be given to determine reflexes. Subjects will also have magnetic resonance imaging(MRI)scans of the cervical spine (neck). Women of child-bearing potential will need to have a urine pregnancy test immediately prior to the MRI scan. Mri scan will take approximately 60 minutes to complete. The clinical examinations will take approximately 30 minutes to complete. Subject participation in this study will be complete following the MRI and clinical examinations.
  Interventions: Other: MRI; Other: Clinical Exam
- Healthy controls (MRI) (Active Comparator): Subjects will also have magnetic resonance imaging (MRI) scans of the cervical spine(neck). Women of child-bearing potential will need to have a urine pregnancy test immediately prior to the MRI scan. Mri scan will take approximately 60 minutes to complete. Subject participation in this study will be complete following the MRI.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Subjects will have magnetic resonance imaging(MRI)scans of the cervical spine(neck). This involves lying on a table and sliding into a scanner consisting of a large magnet. This will take approximately one hour to complete. All subjects will be instructed to remove all jewelry and other metal-containing objects for the scan. During the MRI scan loud noises may be heard. Subjects may have a soft brace for the neck for positioning purposes.
Other: Clinical Exam — Brief neurological exam will be performed.
  Arms: Amyotrophic Lateral Sclerosis

SUMMARY:
The investigators want to know if magnetic resonance imaging can accurately provide an early diagnosis of amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
Currently there is no definitive diagnostic test for amyotrophic lateral sclerosis (ALS). The investigators' goal is to determine if magnetic resonance imaging can provide an accurate diagnosis of ALS by looking at chemical concentrations in the spinal cord at the neck level which show up in MRI imaging and compare these chemical concentrations to corresponding measures in healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 80 years of age.

Exclusion Criteria:

1. Do not have active substance abuse
2. Do not have co-morbid psychiatric disease
3. Do not have opportunistic central nervous system infection
4. Do not have cerebrovascular disease
5. Do not have a contraindication for magnetic resonance imaging(MRI)(e.g. cardiac pacemaker, ferromagnetic or metallic implants).
6. Are not pregnant
7. Have not had cervical spinal surgery(neck) -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Study levels of N-acetylaspartate (NAA)in the cervical spinal cord. | 60 minutes or as needed (rarely more than 2 hours)
  1. Study investigators will measure the differences in the spinal cord metabolite, N-acetylaspartate in ALS subjects compared to healthy controls using magnetic spectroscopy.

SECONDARY OUTCOMES:
Fractional anisotropy in the cervical spinal cord | 3 years
  Study fractional anisotropy levels (unitless) using diffusion tensor imaging in ALS patients compared to healthy controls in the cervical spinal cord.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Foerster, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No